CLINICAL TRIAL: NCT03978351
Title: The Role of Midkine in Diagnosis of Thyroid Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Hassan Thabet Ahmed, Principal investigator, Assiut University
Other Study IDs: Marwa Hassan
Record Dates: First submitted 2018-11-24; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2018-09

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Evaluation of the role of serum midkine in differentiating malignant from benign thyroid nodule
2. studying the level of serum midkine in relation to different thyroid cancer stages

ELIGIBILITY:
Inclusion Criteria:

patient with thyroid nodule

Exclusion Criteria:

1. Other known organ tumour
2. Chemothyrapy
3. Radiothyrapy c. Sample Size Calculation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted on 85 informed and consented individuals (according to the guidelines of ethical committee of faculty of Medicine, Assuit University ) The study will include 30 patients with thyroid cancer and 30 patients with benign thyroid diseases. The study will also include 25 aged matched apparently healthy individuals as a control group.
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
serum midkine levels | Baseline